CLINICAL TRIAL: NCT02803268
Title: A Study to Investigate the Safety, Tolerability and Pharmacokinetics of Multiple Doses of MT-8554 in Female Subjects Experiencing Vasomotor Symptoms
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MT-8554-E04
Record Dates: First submitted 2016-06-14; First posted 2016-06-16 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Vasomotor Symptoms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- MT-8554 low dose (Experimental): Patients who meet eligibility criteria will be administered once daily either low dose of MT-8554 or a matching Placebo from Day 1 to 14.
  Interventions: Drug: MT-8554 low dose; Drug: Placebo
- MT-8554 middle dose (Experimental): Patients who meet eligibility criteria will be administered once daily either middle dose of MT-8554 or a matching Placebo from Day 1 to 14.
  Interventions: Drug: MT-8554 middle dose; Drug: Placebo
- MT-8554 high dose (Experimental): Patients who meet eligibility criteria will be administered once daily either high dose of MT-8554 or a matching Placebo from Day 1 to 14.
  Interventions: Drug: MT-8554 high dose; Drug: Placebo

INTERVENTIONS:
Drug: MT-8554 low dose
  Arms: MT-8554 low dose
Drug: MT-8554 middle dose
  Arms: MT-8554 middle dose
Drug: MT-8554 high dose
  Arms: MT-8554 high dose
Drug: Placebo

SUMMARY:
A Study to Investigate the Safety, Tolerability and Pharmacokinetics of Multiple Doses of MT-8554 in Female Subjects Experiencing Vasomotor Symptoms

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet one of the following criteria:Woman aged ≥18 years with histologically proven non-metastatic breast cancer (Stages I, II or III) and without evidence of disease / Woman aged ≥40 years who are post-menopausal / Woman aged ≥40 years who are peri-menopausal
* Subjects who have ≥7 Vasomotor Symptoms per day on average
* A body weight of ≥45 kg

Exclusion Criteria:

* Participation in more than three clinical studies involving administration of an unlicensed Investigational Medicinal Product in the previous year, or any study within 12 weeks
* Clinically significant endocrine, thyroid, hepatic, respiratory, gastro-intestinal, renal, cardiovascular disease, or history of any significant psychiatric/psychotic illness disorder
* Clinically relevant abnormal medical history, physical findings or laboratory values

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-06; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability as measured by vital signs | Up to Day 21
Safety and Tolerability as measured by number of participants with adverse events | Up to Day 21

SECONDARY OUTCOMES:
Plasma concentration of MT-8554 after dosing | Up to Day 15
Change from baseline in core body temperature | Up to Day 14
Frequency of Vasomotor Symptoms | Up to Day 15

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational center, City Name, Germany